CLINICAL TRIAL: NCT00394784
Title: Surveillance Study - Incidence of Antibiotic Resistance in Serial Gram-negative Bloodstream Isolates
Status: Withdrawn | Type: Observational
Why Stopped: Study terminated due to no enrollment.
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Brian Potoski, Pharm D, University of Pittsburgh
Other Study IDs: IRB0608120
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Gram-negative Bacterial Infections
Keywords: gram negative bacteria; culture; infection
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research is important because it allows for the determination of resistance rates to antibiotics that may not be frequently tested by the clinical microbiology laboratory at University of Pittsburgh Medical Center (UPMC)-Presbyterian. It also will provide antibiotic minimum inhibitory concentrations (MICs) for these pathogens which may help in identifying the best empiric antibiotic option for gram-negative blood stream infections based on known pharmacodynamic parameters.

DETAILED DESCRIPTION:
Bacterial cultures will be ordered in the normal clinical course of the management of patients in the liver transplant ICU by the medical team. These cultures are then processed by the clinical Microbiology laboratory in the normal manner. If these cultures grow a Gram-negative bacteria, they are eligible for this study. Typically the clinical Microbiology laboratory saves these bacteria for a period of time after the final microbiology report. At this time, unless asked otherwise, the bacteria will be placed in biohazardous waste containers for proper disposal. If these cultures have grown a Gram-negative bacteria, they are eligible for this study, and will not be disposed of but will be given to the investigators without identifiers for this study. The antibiotic susceptibility of these organisms will be tested by the investigators in a separate research laboratory. Mechanisms of antibiotic resistance may also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive gram-negative bacteria

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: positive gram negative bacteria isolates
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: Brian Potoski, PharmD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States